CLINICAL TRIAL: NCT03413761
Title: Antioxidant Supplements, Genetics and Chemotherapy Outcomes
Status: Completed | Type: Observational
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: EPR 43304
Record Dates: First submitted 2018-01-05; First posted 2018-01-29 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Node Positive Breast Cancer; Node Negative Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will investigate the null hypothesis that use of antioxidant supplements during adjuvant chemotherapy will have no impact on toxicities and disease-free, as well as overall, survival, and also evaluate the role of polymorphisms in genes related to oxidative stress in relation to treatment outcomes.

DETAILED DESCRIPTION:
This study will enroll 3000 women from S0221with node positive or high-risk node-negative breast cancer receiving AC+T onto this ancillary study to address the following specific aims:

1. To characterize use of antioxidant supplements with a survey instrument prior to and at completion of treatment, and to evaluate reported use pre and post treatment in relation to toxicity and disease-free survival. The potential effects of diet, physical activity, and other lifestyle factors on relationships between supplement use and treatment outcomes will also be considered.
2. To evaluate if variants (polymorphisms) in genes that produce reactive oxygen species (ROS) (MPO) and in genes that protect cells from the effects of ROS are associated with treatment-related toxicities and with disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of operable Stage 1, II, or III invasive breast cancer with known estrogen or progesterone receptor status
* high risk by meeting at least one of the following criteria:

  1. tumor >= 2 cm in greatest diameter
  2. one or more axillary or intramammary nodes are involved by metastatic breast cancer
* had either a modified radical mastectomy or local excision of all tumors plus axillary node dissection or sentinel node resection
* not received prior chemotherapy or radiation therapy for the current malignancy
* no history of congestive heart failure or angina pectoris
* normal creatinine and bilirubin, alkaline phosphatase and SGOT or SGPT 2 x the institutional upper limits of normal
* ANC greater than or equal to 1,200 ul and platelet count of greater than or equal 100,000 U1
* No previous malignancies
* Age 18 or greater
* Performance status of 0 -2 by Zubrod criteria
* HIV negative (if known)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Woman from SWOG trial S0221 with node-positive or high-risk node-negative breast cancer.
Sampling Method: Probability Sample
Enrollment: 1771 (Actual)
Dates: Start 2004-12-18 (Actual); Primary Completion 2013-11-12 (Actual); Study Completion 2013-11-12 (Actual)

PRIMARY OUTCOMES:
Epidemiologic Questionnaire | At baseline interview
  Self administered questionnaire to evaluate use of antioxidant supplements in relation to toxicity
Evaluate if variants in genes are associate with treatment related toxicities | Prior to treatment
  Polymorphisms will be determined by sequencing as described in detail on the National Cancer Institute'sSNP500Cancer database
Evaluate if variants in genes are associate with treatment related toxicities | Year 5
  Polymorphisms will be determined by sequencing as described in detail on the National Cancer Institute'sSNP500Cancer database
Epidemiologic Questionnaire | every 6 months for 5 years
  Self administered questionnaire to evaluate use of antioxidant supplements in relation to disease free survival

REFERENCES:
- [Derived] Mongiovi JM, Zirpoli GR, Cannioto R, Sucheston-Campbell LE, Hershman DL, Unger JM, Moore HCF, Stewart JA, Isaacs C, Hobday TJ, Salim M, Hortobagyi GN, Gralow JR, Thomas Budd G, Albain KS, Ambrosone CB, McCann SE. Associations between self-reported diet during treatment and chemotherapy-induced peripheral neuropathy in a cooperative group trial (S0221). Breast Cancer Res. 2018 Nov 28;20(1):146. doi: 10.1186/s13058-018-1077-9. PMID 30486865